CLINICAL TRIAL: NCT05439668
Title: Comparison of Two Abdominal Exercise Programs on the Interrect Distance in Postpartum Woman
Brief Title: Comparison of Two Abdominal Exercise Programs on the Interrect Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Iria Da Cuña Carrera, Principal investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17062022
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Postpartum Period
Keywords: Abdominal muscle; Interrectus distance; Abdominal hypopressive exercise; Abdominal crunch exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic abdominal exercises Group (Experimental): This group will carry out an abdominal strengthening exercise program based on the classic abdominal exercises.
  Interventions: Other: Classic abdominal strengthening exercises
- Abdominal hypopresives exercise Group (Experimental): This group will carry out an abdominal strengthening exercise program based on the abdominal hypopressives exercises.
  Interventions: Other: Hypopressive abdominal exercises program

INTERVENTIONS:
Other: Classic abdominal strengthening exercises — Classic abdominal strengthening exercises (Curl-up, sit-ups and leg-rise), balance exercises, general mobility and upper limb strengthening exercises.
  Arms: Classic abdominal exercises Group
Other: Hypopressive abdominal exercises program — Hypopressive abdominal exercises, balance exercises, general mobility and upper limb strengthening exercises
  Arms: Abdominal hypopresives exercise Group

SUMMARY:
The objective of the research is to compare two programs of exercises in postpartum woman, one based in abdominal strengthening exercises and the other based in abdominal hypopresive exercise.

DETAILED DESCRIPTION:
Diastasis recti abdominisis the separation of the two rectus abdominis muscles along the linea alba with a consequent separation of fibres and widening of the same. The linea alba has different functions which include supporting the proximal anterior recti, guaranteeing the stability of the vertebral column, pelvis and the pelvic floor, and intervening in the function of the abdominal muscles since it serves as their anterior anchorage.

The crunch abdominal exercise (classic abdominal) is the most studied exercise used to test the behaviour of the linea alba, and in most cases, a decrease in the inter-rectus distance is observed when compared to the resting stage. In the oder hand, Abdominal hypopresives exercises were designed for women in the postpartum period but the effects over the abdominal muscles is unknown and the authors are unaware of any study that evaluates the effect of a hypopressive exercise program on the interrectus distance.

The objective of the research is to compare two programs of exercises in postpartum woman, one based in abdominal strengthening exercises and the other based in abdominal hypopresive exercise.

ELIGIBILITY:
Inclusion Criteria:

* Women having given birth 8 weeks before starting the study treatment
* Women agree to participate in the study
* Women with vaginal delivery.

Exclusion Criteria:

* Women with abdominal hernia
* Pregnancy woman
* Previus Abdominal Surgery

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Interrectus distance measure | Baseline, preintervention
  he participants will be placed in supine decubitus with the knees flexed to 90º with the feet resting on the stretcher and the arms along the body. After receiving the instructions to perform an abdominal crunch, subjects are asked to lift their heads and lift shoulders until the scapula lifts off the table. The ultrasound images will be recorded with an ultrasound scanner (GE Logic and; 4 12MHz, 39mm linear transducer; mode B), in a position of supine rest and a position of muscle activation (isometric contraction), 2 cm and 5 cm above the navel. Centimeters are the unit of measurement.
Interrectus distance measure | After the intervention
  he participants will be placed in supine decubitus with the knees flexed to 90º with the feet resting on the stretcher and the arms along the body. After receiving the instructions to perform an abdominal crunch, subjects are asked to lift their heads and lift shoulders until the scapula lifts off the table. The ultrasound images will be recorded with an ultrasound scanner (GE Logic and; 4 12MHz, 39mm linear transducer; mode B), in a position of supine rest and a position of muscle activation (isometric contraction), 2 cm and 5 cm above the navel. Centimeters are the unit of this measurement.

SECONDARY OUTCOMES:
Maternal age | Preintervention
  Age when the woman gave birth. This variable will be managed by the midwives through their clinical history. Years are the unit of this measurement.
Fetal weight | Preintervenrion
  Weight baby This variable will be managed by the midwives through their clinical history. Kilogrames are the unit of this measurement.
Number of deliveries | Preintervention
  Total of number of deliveries. This variable will be managed by the midwives through their clinical history. Absolut number are the unit of this measurement.
Weight gain during pregnancy | Preintervention
  Weight gain during pregnancy. This variable will be managed by the midwives through their clinical history. Kilogrames are the unit of this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Iria Da Cuña-carrera, PHD, Principal Investigator — Universitu of Vigo
Locations (1):
- Iria Da Cuña Carrera, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Da Cuna-Carrera I, Alonso-Calvete A, Soto-Gonzalez M, Lantaron-Caeiro EM. How Do the Abdominal Muscles Change during Hypopressive Exercise? Medicina (Kaunas). 2021 Jul 9;57(7):702. doi: 10.3390/medicina57070702. PMID 34356983
- [Background] Carrera Perez C, Da Cuna Carrera I, Gonzalez Gonzalez Y. [What is the best exercise for rehabilitation of abdominal diastasis rehabilitation?]. Rehabilitacion (Madr). 2019 Jul-Sep;53(3):198-210. doi: 10.1016/j.rh.2018.12.004. Epub 2019 Apr 11. Spanish. PMID 31370947
- [Background] Da Cuna-Carrera I, Alonso-Calvete A, Lantaron-Caeiro EM, Soto-Gonzalez M. Are There Any Differences in Abdominal Activation between Women and Men during Hypopressive Exercises? Int J Environ Res Public Health. 2021 Jun 29;18(13):6984. doi: 10.3390/ijerph18136984. PMID 34210004
- [Background] Mota P, Pascoal AG, Carita AI, Bo K. The Immediate Effects on Inter-rectus Distance of Abdominal Crunch and Drawing-in Exercises During Pregnancy and the Postpartum Period. J Orthop Sports Phys Ther. 2015 Oct;45(10):781-8. doi: 10.2519/jospt.2015.5459. Epub 2015 Aug 24. PMID 26304639
- [Background] Lee D, Hodges PW. Behavior of the Linea Alba During a Curl-up Task in Diastasis Rectus Abdominis: An Observational Study. J Orthop Sports Phys Ther. 2016 Jul;46(7):580-9. doi: 10.2519/jospt.2016.6536. PMID 27363572
- [Derived] Soto-Gonzalez M, Da Cuna-Carrera I, Lantaron-Caeiro EM, Pascoal AG. Effect of hypopressive and conventional abdominal exercises on postpartum diastasis recti: A randomized controlled trial. PLoS One. 2024 Dec 12;19(12):e0314274. doi: 10.1371/journal.pone.0314274. eCollection 2024. PMID 39666696